CLINICAL TRIAL: NCT07374523
Title: Clinical and Radiographic Evaluation of Local Application of Melatonin on Osseointegration of Immediate Dental Implants for Mandibular Single Rooted Teeth: A Randomized Controlled Study
Brief Title: Clinical and Radiographic Evaluation of Local Application of Melatonin on Osseointegration of Immediate Dental Implants for Mandibular Single Rooted Teeth
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Suez Canal University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1008/2025
Record Dates: First submitted 2026-01-20; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Implant Therapy
Keywords: implant; clinical stability; radiographic assessment; soft tissue health; Melatonin; immediate implant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Melatonin gel (Experimental): implant was placed with melatonin application (3mg Melatonin into 2ml of Hydroxyethyl Cellulose Gel 2%).
  Interventions: Other: Melatonin gel; Other: Control
- control without melatonin gel (Placebo Comparator): implant was placed without melatonin
  Interventions: Other: Melatonin gel; Other: Control

INTERVENTIONS:
Other: Melatonin gel — the implant was placed with melatonin application (3mg Melatonin into 2ml of Hydroxyethyl Cellulose Gel 2%).
Other: Control — the implant was placed without melatonin.

SUMMARY:
Clinical and Radiographic Evaluation of Local Application of Melatonin on Osseointegration of Immediate Dental Implants for Mandibular Single Rooted Teeth:

A Randomized Controlled Study

DETAILED DESCRIPTION:
Dental implant is a treatment option that offers great functional and biologic advantages alongside noticeable long-term success outcomes with survival rates exceeding 95% . Delayed implant placement has been widely and successfully used for replacing missing teeth However, there are some challenges faced with delayed implant placement protocol due to the postextraction alveolar ridge resorption in buccolingual and apicocoronal directions .

The percentage of the post-extraction horizontal and vertical dimensional changes are 29-63% and 11-22% respectively . This is attributed to the disruption of vascular supply due to damage of periodontal ligament leading to pronounced bundle bone resorption . This pronounced post-extraction bone resorption usually leads to functional challenges and the need for augmentation procedures . In order to avoid such challenges, immediate post-extraction implant placement concept was introduced to avoid the bone resorption following tooth extraction and to reduce treatment time . Immediate implant placement showed a high overall implant placement rate reaching 97.1% as reported in the systematic review and 94.9% in the meta-analysis

Although immediate implant placement is effective in preservation of the alveolar bone dimensions but it fails to completely prevent the postextraction dimensional changes . Therefore, attempts were done regarding placement of various biomaterials in the peri-implant gap to increase the immediate implant stability and to minimize or even prevent the post-extraction bone dimensional changes if possible. Multiple materials were successfully used such as bone grafting materials like xenografts , autogenous graftsin addition to the application of bone morphogenetic proteins (BMPs), platelet rich fibrin (PRF) .

Melatonin (MLT) among these agents which are of a great interest for the recent researches whether in the medical or dental fields due to their confirmed physiological and structural functions, their biocompatibility and non-antigenic properties .

MLT is a natural hormone with powerful antioxidant properties, released mainly the pineal gland . It is successfully used in various conditions as sleep disorders, cardiovascular, chronic inflammatory diseases and parkinsonism

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged between 21 and 60 years.
2. Good general health (ASA I).
3. Non-smokers or light smokers (<10 cigarettes/day).
4. Presence of a single non-restorable mandibular tooth indicated for extraction (incisor, canine, or premolar).
5. Adequate bone volume to receive a dental implant.
6. Patients with good oral hygiene.

Exclusion Criteria:

1. Medically compromised patients (e.g., uncontrolled diabetes, immunosuppressive therapy, bisphosphonate use)
2. Pregnant and lactating women.
3. Active periodontal disease at the implant site.
4. Acute infection at the extraction site (abscess or sinus tract).
5. Severe parafunctional habits (e.g., bruxism, clenching).

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2025-09-01 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Implant stability (ISQ) | Immediately postoperatively and at 6months postoperatively
  Implant stability will be evaluated using resonance frequency analysis and recorded as ISQ values at the specified time points.

SECONDARY OUTCOMES:
post-operative pain (VAS) | At 1, 3 and 7 days postoperatively
  Postoperative pain assessed using visual analogue scale (VAS)
  Visual Analog Scale (VAS) for Pain, Grades:
  0 - No pain 1-3 - Mild pain (nagging, annoying, but not interfering with activities) 4-6 - Moderate pain (interferes significantly with activities) 7-10 - Severe pain (disabling, unable to perform activities)
post-operative Edema | At 1, 3 and 7 days postoperatively
  Post-operative Edema Scale (Grade 0-3) Grades:
  Grade 0: No edema observed Grade 1: Intraoral edema only Grade 2: Extraoral edema Grade 3: Diffuse edema involving both intraoral and extraoral areas
Marginal bone loss | Each patient will be radiographically assessed immediately postoperative, after 3 months and after 6 months.
  Marginal bone loss:
  measured using DIGORA software (Soredex, Helsinki, Finland) by calculating the vertical distance (in mm) from the implant shoulder/platform to the first bone-to-implant contact on mesial and distal aspects.
Bone density | Each patient will be radiographically assessed immediately postoperative, after 3 months and after 6 months.
  bone density around each implant will be assessed using DIGORA software (Soredex, Helsinki, Finland).
  A standardized region of interest (ROI) will be selected adjacent to the implant, and the mean gray scale values will be calculated to represent bone density.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry Suez Canal University, Ismailia, Egypt, Egypt